CLINICAL TRIAL: NCT05986188
Title: Evaluating a School-based Social and Material Needs Identification System to Prevent Youth Violence Involvement
Status: Active, not recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Wayne State University (Other); The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Rebeccah Sokol, Assistant Professor, School of Social Work, University of Michigan
Other Study IDs: R01CE003536 (NIH)
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-08

CONDITIONS: Violence, Physical; Maltreatment, Child
Keywords: material needs; social needs; intervention; school-based; school violence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Implementing Schools: Implementing schools are public K-12 schools in the State of Michigan that participated in the Pathways to Potential program in a given year (from 2012 to 2024).
  Interventions: Other: Pathways to Potential
- Non-implementing schools: Non-implementing schools are public K-12 schools in the State of Michigan that DID NOT participate in the Pathways to Potential program in a given year (from 2012 to 2024).

INTERVENTIONS:
Other: Pathways to Potential — Pathways to Potential stations MDHHS caseworkers, called success coaches, in local elementary, middle, and high schools. After identifying a social or material need that is a barrier to school attendance (e.g., transportation barriers, caregiver unemployment), success coaches connect students and families to community resources and public assistance.
  Groups: Implementing Schools

SUMMARY:
The goal of this observational study is to evaluate the effects of Pathways to Potential (P2P) on youth violence involvement in Michigan public K-12 students. The main goals of this study are:

* This project will link longitudinal P2P participation data to state administrative records and school disciplinary data to evaluate associations between school P2P participation and youth outcomes-specifically chronic absenteeism, peer aggression expulsions, and child maltreatment rates within a school (Aim 1).
* Given the focus of P2P is to improve the social and structural conditions within a school that contribute to student chronic absenteeism, the team will assess if chronic absenteeism rates mediate the relationships between school P2P participation and youth violence involvement (Aim 2).
* Finally, a survey of success coaches will inform the examination of school and implementation factors that moderate associations between P2P participation and youth violence involvement (Aim 3).

Schools participating in P2P receive Michigan Department of Health and Human Services (MDHHS) caseworkers, called success coaches, in local elementary, middle, and high schools. After identifying a social or material need that is a barrier to school attendance (e.g., transportation barriers, caregiver unemployment), success coaches connect students and families to community resources and public assistance.

ELIGIBILITY:
Administrative Data Inclusion Criteria:

* State of Michigan K-12 public school
* In person instruction
* Open to all students in District/area

Administrative Data Exclusion Criteria:

* Private schools
* Virtual learning
* Needs-specific schools

Survey Inclusion Criteria:

* 18 years of age and older
* Working as a Success Coach inside a Michigan K-12 public school during the data collection period

Survey Exclusion Criteria:

* Former Success Coaches
* Success Coaches not working inside a Michigan K-12 public school during the data collection period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Almost all of the data used for analyses will come from secondary administrative datasets acquired through Data Use Agreements with specific State of Michigan agencies (i.e. Michigan Department of Health and Human Services and the Michigan Department of Education).
  The survey portion of this study will ONLY be administered to Success Coaches over the age of 18 who are actively working inside of a K-12 public school at the time of the collection period.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Peer aggression expulsions | Peer aggression expulsions will be measured for every academic school year from 2001 to 2022, possibly to 2024 depending on data availability
  The state of Michigan requires all public schools to report expulsions for all students to the Michigan Department of Education (MDE), including the incident type(s) which led to the expulsion. Expulsions are instances in which the local educational agency removes a student from their regular school for disciplinary purposes for the remainder of the school year or longer. The investigators will consider expulsions for peer aggression as expulsions which included any of the following: 1) firearm possession-handgun; 2) firearm possession-rifle/shotgun; 3) firearm possession-other firearm; 4) other weapon possession; 5) bomb or similar threat; 6) arson; 7) physical violence with injury, or; 8) physical violence without injury. For each school, the study team will calculate the total number of peer aggression expulsions per school year.
Child maltreatment | Peer aggression expulsions will be measured for every academic school year from 2001 to 2022, possibly to 2024 depending on data availability
  The Michigan Statewide Automated Child Welfare Information System (MiSACWIS) includes dates of investigations into child maltreatment, names of alleged victims, and date of birth of alleged victims for all child maltreatment investigations in the state of Michigan. Investigators will link the MiSACWIS data to individual student data from MDE that includes information on student name, date of birth, schools of enrollment, and dates of school enrollment enrolled schools. The study team will use this linked dataset to calculate the number of child maltreatment investigations per school per school year.
Chronic absenteeism | Chronic absenteeism will measured for every academic school year from 2004 to 2022, possibly to 2024 depending on data availability
  A student is considered chronically absent if they miss 10% or more of school days in which they are enrolled at the school. For each school, the investigators will calculate the total number of students that were chronically absent via the data provided by MDE.

SECONDARY OUTCOMES:
Firearm-involved expulsions | Firearm-involved expulsions will be measured for every academic school year from 2001 to 2022, possibly to 2024 depending on data availability
  In the state of Michigan, firearm possession on school grounds by a student requires the student to be expelled from the school. Expulsions for firearm possession on school grounds can be recorded as one or more of the following incident types: 1) firearm possession-handgun; 2) firearm possession-rifle/shotgun; 3) firearm possession-other firearm. The study team will consider any expulsions that included one of these types as a reason for expulsion as a firearm-involved expulsion. For each school, the study team will calculate the total number of firearm-involved expulsions per school year.

CONTACTS AND LOCATIONS:
Overall Officials: Rebeccah L Sokol, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will not be shared with other researchers.
  MDHHS P2P Data: The Data Use Agreement (DUA) stipulates that the data must only be used by members of the study team and that it must be destroyed at the conclusion of the study.
  MDE K-12 Data: This dataset contains Personally Identifiable Information individual-level student data protected under FERPA. The dataset cannot be made publicly available without violating FERPA regulations, risking deductive disclosure, or violating the DUA.
  MDHHS MiSACWIS Data: This dataset contains Personally Identifiable Information and sensitive details about child maltreatment investigations. The data cannot be made publicly available without risking deductive disclosure or violating the DUA.
  Success Coach Survey data: The survey data will be deidentified and stored in the University of Michigan's Inter-University Consortium for Political and Social Research's (ICPSR) OpenICPSR repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available within a year of the collection completion data (June 2025) and will remain available indefinitely.
Access Criteria: Researchers will be able to access individual level, anonymized success coach implementation questionnaire data. Can be found through the openICPSR data repository and accessed by creating a free account (https://doi.org/10.3886/E236862V1).
URL: https://www.openicpsr.org/openicpsr/about

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT05986188/Prot_SAP_001.pdf